CLINICAL TRIAL: NCT04906915
Title: Effect of Ketamine Assisted Analgesia on Oxygen Supply and Oxygen Consumption in Patients After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Xingui Dai, Critical Care Medicine, First People's Hospital of Chenzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ketamine
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Intensive Care Unit
Keywords: Ketamine; Extracorporeal circulation; Oxygen Supply; Oxygen Consumption
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): The experimental group was continuously pumped with remifentanil + ketamine for analgesia, and the control group was continuously pumped with remifentanil + placebo (normal saline) for analgesia. RASS and CPOT scores were performed to evaluate the pain degree of the patients.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — The efficacy of ketamine was assessed by calculating oxygen supply and consumption

SUMMARY:
After cardiopulmonary bypass heart surgery, with the rewarming of body temperature, the metabolic capacity of the body is enhanced, the microcirculation is opened, and tissue perfusion is increased. At the same time, the body pays off the oxygen debt formed by the low temperature and reduced blood flow in cardiopulmonary bypass, so that the tissue oxygen demand increases and oxygen consumption increases.Analgesia and sedation are important treatment measures for patients after cardiopulmonary bypass. S-isomer of ketamine and eselamine enhanced the sedation and enhanced the analgesic effect, but whether it can improve the imbalance of oxygen supply and oxygen consumption after cardiopulmonary bypass is unknown.

DETAILED DESCRIPTION:
After cardiopulmonary bypass, the body usually appears in a state of hypermetabolism. In addition to anesthesia resuscitation and recovery of spontaneous respiration, chills, pain and anxiety can increase oxygen demand, increased oxygen consumption is also related to a series of neuroendocrine reactions.At the same time, the body needs to repay the oxygen debt formed by low temperature and reduced blood flow in extracorporeal circulation, so that the tissue oxygen demand increases, and the systemic oxygen consumption is significantly higher than the normal physiological state.

Sedation and analgesia treatment is one of the important early treatment measures for patients after heart surgery. Patients with heart disease are prone to anxiety and restlessness due to reduced cardiac function reserve, severe surgical trauma and extracorporeal circulation, which can lead to hemodilution, tissue edema, ischemia and reperfusion injury, etc. In addition, patients with high preoperative mental stress are prone to anxiety and restlessness.Appropriate sedation and analgesia treatment is very important to reduce stress response, reduce oxygen consumption and maintain the stability of hemodynamics.

The application of ketamine in sedation and analgesia has the characteristics of high controllability, and it does not inhibit respiration and mildly excites circulation, but whether it can improve the imbalance of oxygen supply and demand in patients after cardiopulmonary bypass is unknown.Therefore, it is of great significance to investigate the effect of ketamine on oxygen supply and oxygen consumption of patients after cardiopulmonary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (>18years)patients after heart surgery

Exclusion Criteria:

* Chronic kidney disease (CKD); ECMO or IABP assistance is required; Malignant tumor; Acquired immunodeficiency syndrome; receive psychiatric medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-05-08 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Oxygen Supply and Oxygen Consumption | 0-48 hours
  After the patient was admitted to ICU, femoral artery puncture and catheterization were performed to establish PICCO connection access. At 0h, 4h, 8h, 12h, 16h, 20h, 24h, 32h, 40h and 48h after surgery, ice saline injection was used to measure CO, and central vein and peripheral blood samples were collected for blood gas examination.According to the formula, the patient's oxygen supply and oxygen consumption were calculated: DO2=CO×CaO2×10;CaO2 = 1.34 * SaO2 + 0.003 * Hb PaO2;VO2 = CI x (CaO2 - CvO2).

CONTACTS AND LOCATIONS:
Overall Officials: Dixian DX Luo, MS, Study Director — Chenzhou First People Hospital
Locations (1):
- First Hospital Chenzhou, Chenzhou, Hunan, China